CLINICAL TRIAL: NCT03966833
Title: Using Group Interpersonal Psychotherapy to Improve the Well-Being of Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Berk Ozler, The World Bank (Unknown)
Responsible Party: Principal Investigator, Sarah Baird, Associate Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMU/BRAC 2019
Record Dates: First submitted 2019-05-21; First posted 2019-05-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Mental Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Masking Description: Enumerators will be masked to the treatment assignment of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group-based interpersonal therapy (IPT-G) (Experimental): 14 weeks of group-based interpersonal therapy (IPT-G): StrongMinds is focused on treating depression in Uganda by training community members (in this case ELA club mentors) to act as mentors in IPT-G techniques. This intervention will be offered to 13-19 year old young women who score a 10 or higher on the PHQ-8. These adolescents who take up the offer will then be enrolled in the 14 weeks of therapy. Group therapy sessions build bonds between young women and encourage them to actively engage in the healing process and to support each other in the exploration of their depression triggers. With new healthier patterns and skills, women can learn to manage their current depression and ensure future depressive episodes can be quickly identified and resolved before the onset of any long-term consequences.
  Interventions: Behavioral: IPT-G
- IPT-G + Unconditional Cash Transfer: (Experimental): A one time lump sum of 200,000 UGX (~$54) be provided to all study participants in a random sub-set of intervention (IPT-G) clusters near or at the conclusion of the 14-week therapy. This treatment variation will allow for determination of whether complimentary income support enhances the effects of IPT-G on psychological wellbeing and other outcomes of interest.
  Interventions: Behavioral: IPT-G; Behavioral: Unconditional Cash Transfer
- control (No Intervention): ELA clubs function as normal

INTERVENTIONS:
Behavioral: IPT-G — 14 weeks of group-based interpersonal therapy (IPT-G)
  Arms: IPT-G + Unconditional Cash Transfer:; group-based interpersonal therapy (IPT-G)
Behavioral: Unconditional Cash Transfer — Lump sum cash transfer
  Arms: IPT-G + Unconditional Cash Transfer:

SUMMARY:
Adolescent girls in developing countries face high rates of adversity and are at an elevated risk of depression and other forms of psychological distress. Untreated depression can have negative consequences on life outcomes such as early pregnancies, social exclusion and school dropout. These can result in a cycle of poverty for young women and their families. Despite this being a very pressing problem there is little evidence on what types of interventions can help break the vicious cycle of poor mental health and poverty.

This research program aims to evaluate, through the use of a cluster-Randomized Control Trial (cluster- RCT), the effect of group-based interpersonal psychotherapy (IPT-G) and unconditional cash transfers on adolescent girls' mental health and social functioning. Working with Strong Minds Uganda in collaboration with BRAC Uganda's Empowerment and Livelihood for Adolescents (ELA) clubs, the evidence generated from this research will create a better understanding of whether adolescent mental health improves through this cost-effective approach, and whether improved mental health impacts other outcomes of interest.

ELIGIBILITY:
Inclusion Criteria:

* 13-19 year old female who scores 10 or above on PHQ-8

Exclusion Criteria:

* male
* Score below 10 on PHQ-8

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1914 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Minimal Depression 1a | 6 months
  Score <=10 Primary Health Questionnaire 8 (0-24, higher is worse)
Minimal Depression 1b | 12 months
  Score <=10 Primary Health Questionnaire 8 (0-24, higher is worse)
Minimal Depression 1c | 24 months
  Score <=10 Primary Health Questionnaire 8 (0-24, higher is worse)
Psychological Distress 2a | 6 months
  Score >=3 on the General Health Questionnaire 12 (0-12, higher is worse)
Psychological Distress 2b | 12 months
  Score >=3 on the General Health Questionnaire 12 (0-12, higher is worse)
Psychological Distress 2c | 24 months
  Score >=3 on the General Health Questionnaire 12 (0-12, higher is worse)
Self Esteem a | 6 months
  score on Rosenberg self esteem (0-30, higher is better)
Self Esteem b | 12 months
  score on Rosenberg self esteem (0-30, higher is better)
Self Esteem c | 24 months
  score on Rosenberg self esteem (0-30, higher is better)
Resilience a | 6 months
  score on Child & Youth Resilience Measure-Revised (0-34, higher is better)
Resilience b | 12 months
  score on Child & Youth Resilience Measure-Revised (0-34, higher is better)
Resilience c | 24 months
  score on Child & Youth Resilience Measure-Revised (0-34, higher is better)

SECONDARY OUTCOMES:
Indicator for Self-Reported School Enrollment a | 12 months
  Indicator for enrolled in school (=1 if Adolescent Self-Reports Enrolled in school at time of survey)
Indicator for Self-Reported School Enrollment b | 24 months
  Indicator for enrolled in school (=1 if Adolescent Self-Reports Enrolled in school at time of survey)
incidence of pregnancy a | 12 months
  incidence of pregnancy from baseline
incidence of pregnancy b | 24 months
  incidence of pregnancy from baseline
Child Marriage a | 12 months
  incidence of marriage from baseline
Child Marriage b | 24 months
  incidence of marriage from baseline
Competencies a | 12 months
  Score on competency test. This is a score that takes on a value of 0-3 across a set of three questions on ability to answer skills based math questions. Higher is better
Competencies b | 24 months
  Score on competency test. This is a score that takes on a value of 0-3 across a set of three questions on ability to answer skills based math questions. Higher is better
Indicator for self -reported condom use at last sex a | 12 months
  condom use during last sexual encounter (=1 if Adolescent self reports using a condom at last sex)
indicator for self-reported condom use at last sex b | 24 months
  condom use during last sexual encounter (=1 if Adolescent self reports using a condom at last sex)

CONTACTS AND LOCATIONS:
Locations (1):
- BRAC Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available at the conclusion of the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available at the conclusion of the study.